CLINICAL TRIAL: NCT06685341
Title: A Randomized, Double-Blind, Zolpidem and Placebo-Controlled, 4-Way-Period Crossover, Pharmacokinetics and Pharmacodynamics Study of YZJ-1139 Single-Dose Oral in Healthy Young and Elderly Chinese Subjects
Brief Title: PK/PD Study of YZJ-1139
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: YZJ-1139-1-02
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: Single dose, four-cycle crossover
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Drug: YZJ-1139 high dose group (Experimental): Subjects will be into two groups：Young adult subjects and elderly subjects
  Interventions: Drug: YZJ-1139
- Drug: YZJ-1139 low dose group (Experimental): Subjects will be into two groups：Young adult subjects and elderly subjects
  Interventions: Drug: YZJ-1139
- Drug: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Drug: Zolpidem (Active Comparator)
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: YZJ-1139 — YZJ-1139
  Arms: Drug: YZJ-1139 high dose group; Drug: YZJ-1139 low dose group
Drug: Placebo — Oral tablet
  Arms: Drug: Placebo
Drug: Zolpidem — Oral tablet
  Arms: Drug: Zolpidem

SUMMARY:
Primary Objective： To determine the dose-response relationship of YZJ-1139 in young and elderly Chinese subjects after a single oral administration of different doses, and to compare it with zolpidem at clinical doses.

Secondary Objective: To investigate the safety and tolerability of YZJ-1139 in young and elderly Chinese subjects after a single oral administration of different doses, and to compare it with zolpidem at clinical doses.

ELIGIBILITY:
Inclusion Criteria:

1. Young adults and elderly Chinese healthy subjects, both male and female;
2. Age: [young adult group] 18-45 years old (including the threshold value); [Elderly group]65~75 years old (including the cut-off value);
3. Body weight [only for young adults]: ≥50kg, BMI: 18~28kg/m2 (including the threshold value);
4. Understand and sign the informed consent to participate in the study.

Exclusion Criteria:

1. History of heart, liver, lung, kidney, digestive tract, blood system, neuropsychiatric system and other diseases, including anxiety and depression, that researchers deem clinically significant;
2. Comprehensive physical examination, neurological examination, laboratory examination, ECG examination, etc. indicate that the subject has abnormalities that are judged by the researcher as clinically significant;
3. Poor compliance with the pharmacodynamics training before administration;
4. Have taken any medication in the two weeks prior to study administration, and the investigator judges it may affect the evaluation results;
5. History of food and drug allergy or allergic reaction that the researcher determines to be clinically significant;
6. Serological examination (HBsAg, anti-HCV, anti-HIV, TP-Ab) with positive results;
7. History of alcohol or drug abuse within the year prior to study administration that the investigators believe may have affected the results assessed in this study;
8. Frequent (> 1 time per month) use of hypnotic drugs, and screening and baseline benzodiazepine urine screening positive;
9. Participants who need to work night shifts, stay up late, or stay at least 3 time zones away from the study site within 2 weeks before and during the study;
10. Subjects who could not maintain a regular sleep and rest schedule (get up at 6-8 am and go to sleep at 10-12 PM) within 1 week before and during the study and who were judged by the investigator to be likely to affect the results of this study;
11. Those who could not quit smoking and alcohol drinking as required during the study period or whose carbon monoxide breath test detected >7 ppm during the screening period (further confirmation by urine cotinine test if deemed necessary by the investigators);
12. Participants who have participated in any drug clinical trial as a subject within 3 months prior to study administration;
13. Patients who donated blood or blood products ≥400 mL or 2 units within three months prior to drug administration;
14. Those who do not agree to avoid the use of tobacco, alcohol or caffeinated beverages, or to avoid strenuous exercise, or to avoid other factors affecting the absorption, distribution, metabolism or excretion of drugs within 24 hours before and during the trial;
15. Don't agree or is unable to refrain from eating grapefruit or other related tropical fruits and beverages and from using St. John's Wort during the 24 hours prior to the first dose and during the study period;
16. Women who are pregnant or nursing, or who test positive for serum HCG before trial administration, or who cannot/do not use investigator-approved contraception during the study as required;
17. Those with abnormal cognitive function assessment (MMSE less than 26 points) and judged by the researchers to be clinically significant;
18. Subjects deemed unsuitable for this clinical study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Cmax of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
  Cmax is defined as the maximum concentration of drug
AUCinf of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
  AUCinf is defined as the concentration of drug extrapolated to infinite time
AUClast of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
  AUClast is defined as the concentration of drug from time zero to the last observable concentration
Tmax of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
  Tmax is defined as the time (observed time point) of Cmax
t1/2 of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
CL/F of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
  CL/F is defined as the apparent oral clearance following administration of the drug
Vz/F of YZJ-1139、zolpidem | From Day 1 to Day 2 post single dose；up to 4 weeks
  Vz/F is defined as the apparent volume of distribution of the drug
Left and right saccade peak velocity (SPV) of Eye Movements | From Day 1 to Day 2 post single dose；up to 4 weeks
  Instruct the subject to fix their gaze on the red light spot on the LED display and move their eyes with the light spot. During the test, the head and body must remain still. The test consists of the following two parts, each lasting 2 minutes. Between the two parts, the subject should rest for a certain period of time based on their level of fatigue.
  Part 1: Scanning eye movements Part 2: Smooth pursuit eye movements.
left and right saccade accuracy rate (SacAcc) of Eye Movements | From Day 1 to Day 2 post single dose；up to 4 weeks
  Instruct the subject to fix their gaze on the red light spot on the LED display and move their eyes with the light spot. During the test, the head and body must remain still. The test consists of the following two parts, each lasting 2 minutes. Between the two parts, the subject should rest for a certain period of time based on their level of fatigue.
  Part 1: Scanning eye movements Part 2: Smooth pursuit eye movements.
Left and right saccade eye movement response time (SacRT) of Eye Movements | From Day 1 to Day 2 post single dose；up to 4 weeks
  Instruct the subject to fix their gaze on the red light spot on the LED display and move their eyes with the light spot. During the test, the head and body must remain still. The test consists of the following two parts, each lasting 2 minutes. Between the two parts, the subject should rest for a certain period of time based on their level of fatigue.
  Part 1: Scanning eye movements Part 2: Smooth pursuit eye movements.
Smooth eye movement to the left and right (Smooth) of Eye Movements | From Day 1 to Day 2 post single dose；up to 4 weeks
  Instruct the subject to fix their gaze on the red light spot on the LED display and move their eyes with the light spot. During the test, the head and body must remain still. The test consists of the following two parts, each lasting 2 minutes. Between the two parts, the subject should rest for a certain period of time based on their level of fatigue.
  Part 1: Scanning eye movements Part 2: Smooth pursuit eye movements.
Body Sway | From Day 1 to Day 2 post single dose；up to 4 weeks
  The subject takes off their shoes, spreads their feet shoulder-width apart, and stands on a flat ground 120 cm away from the measuring device. They close their eyes and stand for 2 minutes, and the test measures the body sway amplitude (mm) of the subject during the 2-minute closed-eye period. The test evaluates the subject's postural balance
Simple response time of Choice Reaction Time Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test lasts for 1 minute. During the test, there is a vertical line in the center of the screen. On both sides of the screen, random "left" or "right" words will appear. The participants are required to ignore the word meanings and click the "right" or "left" key based on the word's position.
Simple response accuracy rate of Choice Reaction Time Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test lasts for 1 minute. During the test, there is a vertical line in the center of the screen. On both sides of the screen, random "left" or "right" words will appear. The participants are required to ignore the word meanings and click the "right" or "left" key based on the word's position.
Selective response time of Choice Reaction Time Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  During the test, there was a dividing line in the middle of the screen. During the test, the word "left" or "right" appeared randomly on both sides of the screen. Subjects were asked to ignore the position of the word and click the key "right" or "left" according to the meaning of the word.
Selective response accuracy rate of Choice Reaction Time Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  During the test, there was a dividing line in the middle of the screen. During the test, the word "left" or "right" appeared randomly on both sides of the screen. Subjects were asked to ignore the position of the word and click the key "right" or "left" according to the meaning of the word.
The average reaction time for correct responses of Digit Symbol Substitution Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test time is not more than 2 minutes, the symbol is displayed on the screen, and the subject clicks the corresponding number according to the corresponding relationship between the symbol and the number given below. After clicking or exceeding the upper limit of the reaction time, the subject automatically enters the next symbol.
The number of correct responses of Digit Symbol Substitution Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test time is not more than 2 minutes, the symbol is displayed on the screen, and the subject clicks the corresponding number according to the corresponding relationship between the symbol and the number given below. After clicking or exceeding the upper limit of the reaction time, the subject automatically enters the next symbol.
The average reaction time for incorrect responses of Digit Symbol Substitution Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test time is not more than 2 minutes, the symbol is displayed on the screen, and the subject clicks the corresponding number according to the corresponding relationship between the symbol and the number given below. After clicking or exceeding the upper limit of the reaction time, the subject automatically enters the next symbol.
The number of incorrect responses of Digit Symbol Substitution Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test time is not more than 2 minutes, the symbol is displayed on the screen, and the subject clicks the corresponding number according to the corresponding relationship between the symbol and the number given below. After clicking or exceeding the upper limit of the reaction time, the subject automatically enters the next symbol.
The number of non-responses of Digit Symbol Substitution Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The test time is not more than 2 minutes, the symbol is displayed on the screen, and the subject clicks the corresponding number according to the corresponding relationship between the symbol and the number given below. After clicking or exceeding the upper limit of the reaction time, the subject automatically enters the next symbol.
Immediate recall of Word Recall Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  About 1-2 hours after dosing， First, the subjects were shown 20 unrelated words, each word for a few seconds, and then the subjects were asked to immediately recall the words they just saw.
  The number of correct words in instantaneous recall was recorded respectively
Delayed recall of Word Recall Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  About 1-2 hours later, the subjects were allowed to freely recall the words again, which was delayed recall; The number of correct words in delayed recall was recorded respectively
Delayed recognition of Word Recall Test | From Day 1 to Day 2 post single dose；up to 4 weeks
  The subjects were then presented with 40 words (of which 20 were previously presented words and 20 were confounding words), and were asked to answer one by one whether they were the words they had just seen.
  The number of correct words in delayed extraction was recorded respectively

SECONDARY OUTCOMES:
Adverse events (AEs) | From Day 1 to Day 2 post single dose；up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China